CLINICAL TRIAL: NCT01079572
Title: Cost-Effectiveness of Web-Based Follow Up Following Total Joint Arthroplasty
Brief Title: Cost-Effectiveness of Web-Based Follow Ups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dianne Bryant, Associate Professor, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PSI-2010-01
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Osteoarthritis in the Knee Joint; Osteoarthritis in the Hip Joint
Keywords: osteoarthritis; arthroplasty; web-based; electronic follow-up
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- web-based (Experimental): The patient will undergo xrays at the closest PACs enabled imaging centre and will login and answer questions online. The surgeon will review the images and patient responses and determine whether the patient needs to be seen more urgently or a per routine.
  Interventions: Other: web-based
- in-person (Active Comparator): Patients will attend their follow-up appointments in-person as per usual
  Interventions: Other: in-person

INTERVENTIONS:
Other: in-person — Follow-up appointments will be completed in-person as per usual
  Arms: in-person
Other: web-based — Patients who are at least 2 years following knee or hip replacement will complete a questionnaire online and routine x-rays at a PACS enabled imaging center. The patient's surgeon will receive an email from the database summarizing the patient's responses to key questions and will review the x-rays. The surgeon will determine whether the patient needs to be seen in-person.
  Arms: web-based

SUMMARY:
Complications following total joint arthroplasty are rare, and the majority of follow-up visits are routine. The technology now exists to conduct annual follow-up assessments without having to physically see the patient.

This study will investigate the cost-effectiveness of web-based follow-up assessments compared to standard in-clinic follow-ups. We will also assess patient satisfaction, preference, and the validity of the web-based follow up assessments. Patients coming up to their 1 year follow-up or greater will be randomized to either the web-based group or the usual care group.

Web-based patients will complete all questionnaires using an online database system, and have their x-ray taken at their local radiology facility. The surgeon will review radiographs online. If there are any concerns with the x-ray or responses to questionnaires, arrangements will be made for the patient to be seen at the clinic. Patients in the Usual Care group will come into the clinic for their follow-up assessment and have their x-ray taken at University Hospital as usual.

Online assessment could significantly decrease wait times in orthopaedic clinics, as well as increase availability for OR time and new consultations. This approach could also potentially reduce patient burden by decreasing travel distances, financial burden and time requirements.

ELIGIBILITY:
Inclusion Criteria:

* patients who have had a primary total hip or total knee arthroplasty

Exclusion Criteria:

* patients with osteolysis, or previous complications from their joint replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness | one year

SECONDARY OUTCOMES:
Harris Hip Score | one year
Western Ontario and McMaster Osteoarthritis Index (WOMAC) | one year
SF-12 | one year
Adverse events | one year

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada

REFERENCES:
- [Derived] Marsh J, Hoch JS, Bryant D, MacDonald SJ, Naudie D, McCalden R, Howard J, Bourne R, McAuley J. Economic evaluation of web-based compared with in-person follow-up after total joint arthroplasty. J Bone Joint Surg Am. 2014 Nov 19;96(22):1910-6. doi: 10.2106/JBJS.M.01558. PMID 25410510
- [Derived] Marsh JD, Bryant DM, MacDonald SJ, Naudie DD, McCalden RW, Howard JL, Bourne RB, McAuley JP. Feasibility, effectiveness and costs associated with a web-based follow-up assessment following total joint arthroplasty. J Arthroplasty. 2014 Sep;29(9):1723-8. doi: 10.1016/j.arth.2014.04.003. Epub 2014 Apr 13. PMID 24881023
- [Derived] Marsh J, Bryant D, MacDonald SJ, Naudie D, Remtulla A, McCalden R, Howard J, Bourne R, McAuley J. Are patients satisfied with a web-based followup after total joint arthroplasty? Clin Orthop Relat Res. 2014 Jun;472(6):1972-81. doi: 10.1007/s11999-014-3514-0. Epub 2014 Feb 22. PMID 24562873